CLINICAL TRIAL: NCT00480818
Title: An Ascending Multiple Dose Study of the Safety, Pharmacokinetics (PK), and Pharmacodynamics (PD) of SAM-531 Administered Orally to Healthy Young and Elderly Subjects
Brief Title: Study Evaluating the Safety, Pharmacokinetics, and Pharmacodynamics of SAM-531 in Healthy Young and Elderly Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 3193A1-102
Record Dates: First submitted 2007-05-29; First posted 2007-05-31 (Estimated); Last update posted 2007-12-11 (Estimated); Status verified 2007-12

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — SAM-531

INTERVENTIONS:
Drug: SAM-531

SUMMARY:
To assess the safety and tolerability of ascending multiple oral doses of SAM-531, an investigational drug, in healthy young adult and elderly subjects.To assess the pharmacokinetics (PK) and pharmacodynamics (PD) profiles of multiple oral doses of SAM-531 in healthy young adult and elderly subjects.

ELIGIBILITY:
Inclusion criteria :

* Men or women of nonchildbearing potential aged 18 to 45 years
* Elderly men or women aged 65 years and above as of study day 1.
* Body mass index in the range of 18 to 30 kg/m2 and body weight ≥50 kg. Body weight for elderly subjects must be ≥45 kg.

Exclusion criteria:

* Any significant cardiovascular, hepatic, renal, respiratory, gastrointestinal, endocrine, immunologic, dermatologic, hematologic, neurologic, or psychiatric disease.
* Any clinically important deviation from normal limits in physical examination, vital signs, digital 12-lead ECGs, or clinical laboratory test results.
* Tobacco use or the consumption of any caffeine-containing products (e.g., coffee, tea, chocolate, or soda) or alcoholic beverages within 48 hours before study day 1, or grapefruit or grapefruit-containing products 72 hours before study day 1, and until the end of the inpatient confinement period.
* Elderly men or women aged 65 years and above as of study day 1.
* Body mass index in the range of 18 to 30 kg/m2 and body weight ≥50 kg. Body weight for elderly subjects must be ≥45 kg.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80
Dates: Start 2006-09; Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability

SECONDARY OUTCOMES:
Pharmacokinetics and pharmacodynamics

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (1):
- Rennes, France